CLINICAL TRIAL: NCT01890278
Title: Randomized Phase II Trial of Conventional vs IMRT Whole Brain Radiotherapy for Brain Metastases
Brief Title: Phase II Trial of Conventional Versus IMRT Whole Brain Radiotherapy for Brain Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Good Samaritan Hospital Medical Center, New York (Other)
Responsible Party: Principal Investigator, Johnny Kao, Principal Investigator, Good Samaritan Hospital Medical Center, New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-005
Record Dates: First submitted 2013-06-13; First posted 2013-07-01 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Metastatic Brain Cancer
Keywords: Brain Cancer; Metastatic Brain Cancer; IMRT
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole Brain IMRT (Active Comparator): Whole brain radiation therapy delivered via IMRT (37.5 Gy to brain tumor, 30 Gy to the uninvolved brain in 15 fractions), mean dose of less than 18 Gy to scalp.
  Interventions: Radiation: Whole Brain IMRT
- Conventional whole brain RT (Active Comparator): Conventional whole brain radiation therapy (37.5 Gy to the brain tumors and uninvolved brain in 15 fractions).
  Interventions: Radiation: Conventional Whole Brain RT

INTERVENTIONS:
Radiation: Whole Brain IMRT
  Arms: Whole Brain IMRT
Radiation: Conventional Whole Brain RT
  Arms: Conventional whole brain RT

SUMMARY:
In this study the patient will receive either whole brain radiation therapy given by intensity modulated radiation therapy (IMRT) or standard conventional radiation. In IMRT therapy radiation dose to the parts of the brain that do not contain tumors is reduced. This study will look to see if this approach results in less hair loss or fewer memory Problems, as compared to the standard technique. The study will also look at the effectiveness of both techniques in controlling the growth of the tumor.

DETAILED DESCRIPTION:
SCHEMA For Patients with MRI Evidence of Brain Metastasis within 1 Month Prior to Registration

Prior to Treatment Start Confirmation of patient's insurance coverage prior to receiving study-related procedures to e ensure that treatment with IMRT will not be denied.

Radiation Therapy

1. MRI with Fused CT Simulation
2. Neurocognitive Function Testing
3. Quality of Life Assessment

Arm 1 Whole brain radiation therapy delivered via IMRT (37.5 Gy to the brain tumors, 30 Gy to the uninvolved brain in 15 fractions), mean dose of less than 18 Gy to the scalp

Arm 2 Conventional whole brain radiation therapy (37.5 Gy to the brain tumors and uninvolved brain in 15 fractions)

Patient Population: (See Section 3.0 for Eligibility) At least one radiologically diagnosed brain metastasis associated with a histologically proven diagnosis of a nonhematopoietic malignancy. Patients must be classified as RTOG RPA class I or RPA class II

1.0 INTRODUCTION

1.1 Adverse Effects of Whole-Brain Radiotherapy (WBRT)

Whole brain radiotherapy (WBRT) remains the standard treatment approach for patients with multiple brain metastases. WBRT has been shown to achieve rapid palliation of neurological symptoms and improves overall survival compared to corticosteroids alone for patients with multiple brain metastases 1. Additionally, adjuvant WBRT has been shown to improve local control and time to neurocognitive function decline in patients with limited (1 to 4) brain metastases that are treated with surgery or stereotactic radiosurgery 2-4. Despite significant technical advances in radiation delivery and increased survival in tumors that demonstrate sensitivity to systemic therapies, conventional WBRT has not materially changed in the past 50 years 5. Conventional WBRT is generally well tolerated, save for alopecia, fatigue and short-term neurocognitive decline in patients with a short life expectancy (≤ 6 months) 6-8. In a recent randomized trial at MD Anderson, WBRT after SRS increased the risk of neurocognitive decline ≥ 5 points as assessed by the Hopkins Verbal Learning Test at 4 months after treatment compared to SRS alone (49% vs. 23%, p<0.05) 9. In other studies, development of subsequent brain metastases are a significant contributor to cognitive decline 2, 10-11. In long term survivors (≥ 12 months), irreversible neurocognitive decline has been reported in up to 11% of patients treated with conventional WBRT, although this study utilized daily radiation doses ≥3 Gy per day that are no longer in common use 12. The decline in cognitive function assessed by mini mental status examination may take up to 3 years to manifest 2.

Extensive research has investigated methods of improving the efficacy of WBRT. This included increasing the radiation dose, hyperfractionated radiation schedules and combining WBRT with drug therapy 13-16. Currently, the standard WBRT radiation dose schedule is 30 to 37.5 Gy in 10 to 15 fractions. One promising approach to improve local control and survival has been combining WBRT with stereotactic radiosurgery for patients with 1 to 4 metastases 6, 17. An emerging strategy to reduce the toxicity of WBRT is to administer surgery or SRS alone for patients with limited brain metastases 4, 9. Although this results in a higher risk of brain relapse, some of these recurrences can be salvaged with repeat SRS and/or WBRT. For the majority of patients with brain metastases who require WBRT, little research has focused on improving the therapeutic ratio of WBRT by reducing its toxicity 18.

1.2 Rationale for selective targeting of brain metastases in WBRT

In general, radiation oncologists approach patients by selectively targeting the gross tumor plus margin for microscopic extension and setup uncertainty to the prescription dose while administering a lower dose to areas of subclinical risk 19. This strategy is extensively utilized in brain, head and neck, lung, gastrointestinal, breast, gynecologic, hematologic and genitourinary tumors. In many centers, over half of the patients are treated with IMRT to improve dose distributions to increase efficacy and/or reduce toxicity. Despite the critical physiological role played by the uninvolved brain, the reason this paradigm has not been extended to WBRT likely relates to the general poor prognosis of patients with brain metastases with a median survival of 4 months 20. Selectively targeting brain metastases requires more physician, physicist and radiation therapist effort and the investment of increased resources and cost of treatment for this patient population may be unjustified unless the improved dose distribution translates into significant clinical benefit. In the era of accountable care, determining the cost effectiveness of IMRT vs. conventional WBRT is necessary.

The recent identification of long-term survivors of metastatic cancer treated with more effective local and systemic therapies is slowly changing these attitudes 21-22. There are distinct subgroups of patients with brain metastases with a more reasonable prognosis. For instance RTOG recursive partitioning analysis (RPA) group 1 patients have a median survival of 7 months 20. Patients with single brain metastases undergoing surgery followed by WBRT have a median survival of 10 months 4. A recent study from Japan further classified RTOG RPA class II to Class IIa, IIb and IIc based on the presence of favorable factors including performance status, number of brain tumors, primary tumor controlled or active and extracranial metastases 23. Survival for patients with RPA class IIa, IIb and IIc was 16 to 20 months, 8 months and 4 to 5 months respectively with long-term survivors in each subgroup.

There have been preliminary efforts to apply IMRT to improve whole brain radiation. This concept was first proposed by Kao, et al in 2005 24. Two avenues of research were proposed. One approach is to selectively spare parts of the brain that are critical for neurocognitive function, such as the hippocampal stem cells in the subgranular zone 25. This approach has been extensively tested by investigators at the University of Wisconsin. The risk of brain metastases in the hippocampal avoidance zone is less than 5% 26-27. RTOG 0933 is an ongoing phase II trial testing IMRT WBRT to a total dose of 30 Gy in 10 fractions while limiting the mean hippocampal avoidance zone dose to less than 10 Gy 25. The major criticism of this approach is that the hippocampal avoidance zone is only one of several regions of the brain are involved with memory processing and retention 28. Using the RTOG 0933 technique, potentially functional brain tissue including the limbic circuit and neural stem cell region will receive the full prescription dose even if clinically uninvolved with metastases. Pending further study, this approach remains experimental and should not be performed outside the context of controlled clinical trials.

A second strategy is to selectively boost areas of gross disease while simultaneously treating the uninvolved brain with standard radiation doses 24. This strategy is currently being tested in countries with socialized health systems such as the United Kingdom and Canada as a cost-effective alternative to stereotactic radiosurgery boost. A published report from England reported the feasibility of treating gross tumors to 40 Gy in 10 fractions while treating the uninvolved brain to 30 Gy in 10 fractions 29.

A third application of whole brain radiation is selective sparing of the scalp 30. The clinical target is the whole brain but unintended radiation to the scalp can result in temporary or permanent alopecia. Due to the dose distribution of conventional WBRT, the vertex of the scalp receives a particularly high dose. Preliminary work suggests that IMRT can limit the mean scalp dose to 16 to 18 Gy and these reduced doses may shorten the duration of temporary alopecia and possibly reduce the risk of permanent alopecia 30-32.

A final strategy has not yet been explored. Rather than increasing the dose of radiation to the identified brain tumors, we can reduce the dose to the uninvolved brain to reduce acute and long term side effects. In the setting of prophylactic WBRT for small cell and non-small cell lung cancer, lower radiation doses of 25 to 30 Gy in 10 to 15 fractions are considered standard treatment 33-35. In a randomized trial of prophylactic cranial irradiation for small cell lung cancer, there was no evidence of improved disease control with 36 Gy vs. 25 Gy 34. With the exception of a single report demonstrating subtle effects on neurocognitive function as assessed by Hopkins Verbal Learning Test, there is little evidence that WBRT to 25 to 30 Gy in 10 to 15 fractions results in neurocognitive decline with prophylactic WBRT vs. observation in multiple randomized controlled trials 35-36. Higher doses of WBRT have been shown to reduce verbal memory function 37. Additionally, there are robust data from randomized trials reproducibly demonstrating a significant reduction in the incidence of subsequent brain metastases in regions of the brain with no dominant mass appreciable on MRI prior to treatment 33, 35, 38. A theoretical disadvantage of limiting WBRT to 30 Gy in 15 fractions is that this dose may be inadequate to prevent relapse in relatively radioresistant tumors. However, as discussed earlier, some investigators are now administering 0 Gy to uninvolved sites by deferring WBRT due to concerns of toxicity 11.

1.3 Feasibility of Selective Avoidance of Uninvolved Brain and Scalp during IMRT

Based on this body of published evidence, we started utilizing IMRT for selected patients with brain metastases in June 2012. Our planning objectives are to deliver 37.5 Gy in 15 fractions to the gross tumor(s) + 5 mm margin while limiting radiation dose to 30 Gy. A secondary goal is to limit the mean scalp dose to 16 to 18 Gy. No effort was made to achieve additional sparing of the hippocampal stem cells since definitive data demonstrating a benefit has not yet been published. Based on the feasibility and promising preliminary experience, we propose a prospective randomized trial to determine whether there are significant benefits for WBRT delivered via IMRT.

1.4 Neurocognitive Function and Quality of Life Assessment

Although more extensive and sensitive neurocognitive tests such as the Hopkins Verbal Learning Test are available, in the context of resources available to a high-quality community hospital program, we will limit our neurocognitive function assessment to serial mini-mental status examinations. Mini-mental status examination (MMSE) is the most widely used global mental status measure in medical settings and requires less than 10 minutes to complete. This assessment tool has been extensively validated in nearly 2,000 patients with brain tumors treated on RTOG protocols 39.

Quality of life will be assessed using the EORTC QLQ - BN20, which is an extensively validated one page patient-reported survey of 20 questions. The EORTC-QLQ-BN20 is designed for use with patients undergoing chemotherapy or radiotherapy, and is composed of 20 questions assessing visual disorders, motor dysfunction, communication deficit, various disease symptoms (eg, headaches and seizures), treatment toxicities (eg, hair loss), and future uncertainty. The EORTC QLQ - BN20 has robust psychometric properties resulting from rigorous testing, development, and external validity 40.

Within 2 weeks prior to WBRT, all patients will undergo a baseline quality of life assessment.

After completion WBRT, all patients will undergo quality of life assessments every 3 months for 6 months and then every 4 months after whole brain radiotherapy. Quality of life assessments will be scored by a blinded reviewer to avoid potential bias.

1.5 Summary

In summary, preclinical and clinical evidence suggests that radiation dose received by uninvolved portions of the brain during WBRT plays a critical role in causing radiation-induced alopecia and neurocognitive decline without improving survival. Extensive data from randomized trials suggests a benefit in reduced brain relapse from elective treatment of uninvolved brain. Although other approaches are being pursued, reducing the radiation dose to levels utilized for prophylactic cranial irradiation is an attractive alternative to conventional WBRT that non-specifically irradiates the entire brain or eliminating WBRT entirely. We hypothesize that IMRT-WBRT will reduce the incidence and duration of alopecia while reducing the incidence of neurocognitive deficit to the acceptable levels observed in prophylactic cranial irradiation.

ELIGIBILITY:
ELIGIBILITY CHECKLIST

Inclusion Criteria:

* Evidence of at least one brain metastasis on a gadolinium contrast-enhanced MRI
* Pathologic/histological/cytologic proof of a diagnosis of a non-hematopoietic malignancy within 5 years of study entry.
* Patient ≥18 years of age?
* Fall into RTOG Recursive Partition Analysis (RPA) class I or II.
* Karnofsky Performance Score ≥70. (See Appendix III)
* Biopsy done at least 1 week prior to registration. (This requirement does not apply to stereotactic biopsies.)

Exclusion Criteria:

* Contraindication to MR imaging such as implanted metal devices or foreign bodies, severe claustrophobia.
* Creatinine level > 1.4 mg/dl drawn ≤30 days prior to study entry.
* Severe, active co-morbitities.
* Unstable angina, and/or congestive heart failure requiring hospitalization within the last 6 months.
* Transmural myocardial infarction within the last 6 months
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
* Uncontrolled, clinically significant cardiac arrhythmias
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-06; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Alopecia | 1 to 4 months after radiation
  In this study the patient will receive either whole brain radiation therapy given by intensity modulated radiation therapy (IMRT) or standard conventional radiation. In IMRT therapy radiation dose to the parts of the brain that do not contain tumors is reduced.

SECONDARY OUTCOMES:
The study will also look at the effectiveness of both techniques in controlling the growth of the tumor. | 1 year
  IMRT is more expensive than conventional treatment therefor it is important to evaluation whether the newer technique improves quality of life.
Quality of life | 1 year after radiation
  Quality of life as assessed by Mini-mental status examination and patient reported EORTC-BN20 instrument

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Kao, MD, Principal Investigator — Good Samaritan Hospital Medical Center
Locations (1):
- Good Samaritan Hospital Medical Center, West Islip, New York, United States

REFERENCES:
- [Background] Horton J, Baxter DH, Olson KB. The management of metastases to the brain by irradiation and corticosteroids. Am J Roentgenol Radium Ther Nucl Med. 1971 Feb;111(2):334-6. doi: 10.2214/ajr.111.2.334. No abstract available. PMID 5541678
- [Background] Aoyama H, Shirato H, Tago M, Nakagawa K, Toyoda T, Hatano K, Kenjyo M, Oya N, Hirota S, Shioura H, Kunieda E, Inomata T, Hayakawa K, Katoh N, Kobashi G. Stereotactic radiosurgery plus whole-brain radiation therapy vs stereotactic radiosurgery alone for treatment of brain metastases: a randomized controlled trial. JAMA. 2006 Jun 7;295(21):2483-91. doi: 10.1001/jama.295.21.2483. PMID 16757720
- [Background] Kocher M, Soffietti R, Abacioglu U, Villa S, Fauchon F, Baumert BG, Fariselli L, Tzuk-Shina T, Kortmann RD, Carrie C, Ben Hassel M, Kouri M, Valeinis E, van den Berge D, Collette S, Collette L, Mueller RP. Adjuvant whole-brain radiotherapy versus observation after radiosurgery or surgical resection of one to three cerebral metastases: results of the EORTC 22952-26001 study. J Clin Oncol. 2011 Jan 10;29(2):134-41. doi: 10.1200/JCO.2010.30.1655. Epub 2010 Nov 1. PMID 21041710
- [Background] Patchell RA, Tibbs PA, Regine WF, Dempsey RJ, Mohiuddin M, Kryscio RJ, Markesbery WR, Foon KA, Young B. Postoperative radiotherapy in the treatment of single metastases to the brain: a randomized trial. JAMA. 1998 Nov 4;280(17):1485-9. doi: 10.1001/jama.280.17.1485. PMID 9809728
- [Background] Graham PH, Bucci J, Browne L. Randomized comparison of whole brain radiotherapy, 20 Gy in four daily fractions versus 40 Gy in 20 twice-daily fractions, for brain metastases. Int J Radiat Oncol Biol Phys. 2010 Jul 1;77(3):648-54. doi: 10.1016/j.ijrobp.2009.05.032. Epub 2009 Oct 14. PMID 19836153
- [Background] Wong J, Hird A, Kirou-Mauro A, Napolskikh J, Chow E. Quality of life in brain metastases radiation trials: a literature review. Curr Oncol. 2008 Oct;15(5):25-45. doi: 10.3747/co.v15i5.290. PMID 19008990
- [Background] Chang EL, Wefel JS, Hess KR, Allen PK, Lang FF, Kornguth DG, Arbuckle RB, Swint JM, Shiu AS, Maor MH, Meyers CA. Neurocognition in patients with brain metastases treated with radiosurgery or radiosurgery plus whole-brain irradiation: a randomised controlled trial. Lancet Oncol. 2009 Nov;10(11):1037-44. doi: 10.1016/S1470-2045(09)70263-3. Epub 2009 Oct 2. PMID 19801201
- [Background] Li J, Bentzen SM, Renschler M, Mehta MP. Regression after whole-brain radiation therapy for brain metastases correlates with survival and improved neurocognitive function. J Clin Oncol. 2007 Apr 1;25(10):1260-6. doi: 10.1200/JCO.2006.09.2536. PMID 17401015
- [Background] Suh JH. Stereotactic radiosurgery for the management of brain metastases. N Engl J Med. 2010 Mar 25;362(12):1119-27. doi: 10.1056/NEJMct0806951. No abstract available. PMID 20335588
- [Background] DeAngelis LM, Delattre JY, Posner JB. Radiation-induced dementia in patients cured of brain metastases. Neurology. 1989 Jun;39(6):789-96. doi: 10.1212/wnl.39.6.789. PMID 2725874
- [Background] Borgelt B, Gelber R, Kramer S, Brady LW, Chang CH, Davis LW, Perez CA, Hendrickson FR. The palliation of brain metastases: final results of the first two studies by the Radiation Therapy Oncology Group. Int J Radiat Oncol Biol Phys. 1980 Jan;6(1):1-9. doi: 10.1016/0360-3016(80)90195-9. No abstract available. PMID 6154024
- [Background] Knisely JP, Berkey B, Chakravarti A, Yung AW, Curran WJ Jr, Robins HI, Movsas B, Brachman DG, Henderson RH, Mehta MP. A phase III study of conventional radiation therapy plus thalidomide versus conventional radiation therapy for multiple brain metastases (RTOG 0118). Int J Radiat Oncol Biol Phys. 2008 May 1;71(1):79-86. doi: 10.1016/j.ijrobp.2007.09.016. Epub 2007 Dec 31. PMID 18164847
- [Background] Mehta MP, Rodrigus P, Terhaard CH, Rao A, Suh J, Roa W, Souhami L, Bezjak A, Leibenhaut M, Komaki R, Schultz C, Timmerman R, Curran W, Smith J, Phan SC, Miller RA, Renschler MF. Survival and neurologic outcomes in a randomized trial of motexafin gadolinium and whole-brain radiation therapy in brain metastases. J Clin Oncol. 2003 Jul 1;21(13):2529-36. doi: 10.1200/JCO.2003.12.122. PMID 12829672
- [Background] Murray KJ, Scott C, Greenberg HM, Emami B, Seider M, Vora NL, Olson C, Whitton A, Movsas B, Curran W. A randomized phase III study of accelerated hyperfractionation versus standard in patients with unresected brain metastases: a report of the Radiation Therapy Oncology Group (RTOG) 9104. Int J Radiat Oncol Biol Phys. 1997 Oct 1;39(3):571-4. doi: 10.1016/s0360-3016(97)00341-6. PMID 9336134
- [Background] Nieder C. Stereotactic radiosurgery plus whole brain radiotherapy versus radiotherapy alone for patients with multiple brain metastases: regarding Kondziolka et al. IJROBP 1999;45:427-434. Int J Radiat Oncol Biol Phys. 2000 Mar 1;46(4):1081-2. doi: 10.1016/s0360-3016(99)00469-1. No abstract available. PMID 10755878
- [Background] Gondi V, Tome WA, Mehta MP. Why avoid the hippocampus? A comprehensive review. Radiother Oncol. 2010 Dec;97(3):370-6. doi: 10.1016/j.radonc.2010.09.013. Epub 2010 Oct 20. PMID 20970214
- [Background] Kao J, Genden EM, Gupta V, Policarpio EL, Burri RJ, Rivera M, Gurudutt V, Som PM, Teng M, Packer SH. Phase 2 trial of concurrent 5-fluorouracil, hydroxyurea, cetuximab, and hyperfractionated intensity-modulated radiation therapy for locally advanced head and neck cancer. Cancer. 2011 Jan 15;117(2):318-26. doi: 10.1002/cncr.25374. Epub 2010 Sep 9. PMID 20830768
- [Background] Gaspar L, Scott C, Rotman M, Asbell S, Phillips T, Wasserman T, McKenna WG, Byhardt R. Recursive partitioning analysis (RPA) of prognostic factors in three Radiation Therapy Oncology Group (RTOG) brain metastases trials. Int J Radiat Oncol Biol Phys. 1997 Mar 1;37(4):745-51. doi: 10.1016/s0360-3016(96)00619-0. PMID 9128946
- [Background] Kao J, Packer S, Vu HL, Schwartz ME, Sung MW, Stock RG, Lo YC, Huang D, Chen SH, Cesaretti JA. Phase 1 study of concurrent sunitinib and image-guided radiotherapy followed by maintenance sunitinib for patients with oligometastases: acute toxicity and preliminary response. Cancer. 2009 Aug 1;115(15):3571-80. doi: 10.1002/cncr.24412. PMID 19536893
- [Background] Milano MT, Katz AW, Zhang H, Okunieff P. Oligometastases treated with stereotactic body radiotherapy: long-term follow-up of prospective study. Int J Radiat Oncol Biol Phys. 2012 Jul 1;83(3):878-86. doi: 10.1016/j.ijrobp.2011.08.036. Epub 2011 Dec 13. PMID 22172903
- [Background] Yamamoto M, Sato Y, Serizawa T, Kawabe T, Higuchi Y, Nagano O, Barfod BE, Ono J, Kasuya H, Urakawa Y. Subclassification of recursive partitioning analysis Class II patients with brain metastases treated radiosurgically. Int J Radiat Oncol Biol Phys. 2012 Aug 1;83(5):1399-405. doi: 10.1016/j.ijrobp.2011.10.018. Epub 2011 Dec 29. PMID 22209155
- [Background] Knisely JP, Yu JB. Hippocampal-sparing whole-brain radiotherapy: a "how-to" technique using helical tomotherapy and linear accelerator-based intensity-modulated radiotherapy: in regard to Gondi v, et al. (Int j radiat oncol biol phys 2010;78:1244-1252). Int J Radiat Oncol Biol Phys. 2011 Mar 1;79(3):957-8; author reply 958. doi: 10.1016/j.ijrobp.2010.11.001. No abstract available. PMID 21281899
- [Background] Ghia A, Tome WA, Thomas S, Cannon G, Khuntia D, Kuo JS, Mehta MP. Distribution of brain metastases in relation to the hippocampus: implications for neurocognitive functional preservation. Int J Radiat Oncol Biol Phys. 2007 Jul 15;68(4):971-7. doi: 10.1016/j.ijrobp.2007.02.016. Epub 2007 Apr 18. PMID 17446005
- [Background] Marsh JC, Herskovic AM, Gielda BT, Hughes FF, Hoeppner T, Turian J, Abrams RA. Intracranial metastatic disease spares the limbic circuit: a review of 697 metastatic lesions in 107 patients. Int J Radiat Oncol Biol Phys. 2010 Feb 1;76(2):504-12. doi: 10.1016/j.ijrobp.2009.02.038. PMID 20117288
- [Background] Marsh JC, Gielda BT, Herskovic AM, Abrams RA. Cognitive Sparing during the Administration of Whole Brain Radiotherapy and Prophylactic Cranial Irradiation: Current Concepts and Approaches. J Oncol. 2010;2010:198208. doi: 10.1155/2010/198208. Epub 2010 Jun 27. PMID 20671962
- [Background] Edwards AA, Keggin E, Plowman PN. The developing role for intensity-modulated radiation therapy (IMRT) in the non-surgical treatment of brain metastases. Br J Radiol. 2010 Feb;83(986):133-6. doi: 10.1259/bjr/28596848. Epub 2009 Dec 17. PMID 20019176
- [Background] Goffman TE. Permanent alopecia after cranial irradiation: dose-response relationship: in regards to Lawenda et al. (Int J Radiat Oncol Biol Phys 2004;60:879-886). Int J Radiat Oncol Biol Phys. 2005 May 1;62(1):297-8; author reply 298. doi: 10.1016/j.ijrobp.2005.01.048. No abstract available. PMID 15850944
- [Background] Severs GA, Griffin T, Werner-Wasik M. Cicatricial alopecia secondary to radiation therapy: case report and review of the literature. Cutis. 2008 Feb;81(2):147-53. PMID 18441767
- [Background] Gore E. RTOG 0214: a phase III comparison of prophylactic cranial irradiation versus observation in patients with locally advanced non-small cell lung cancer. Clin Adv Hematol Oncol. 2005 Aug;3(8):625-6. No abstract available. PMID 16167048
- [Background] Le Pechoux C, Dunant A, Senan S, Wolfson A, Quoix E, Faivre-Finn C, Ciuleanu T, Arriagada R, Jones R, Wanders R, Lerouge D, Laplanche A; Prophylactic Cranial Irradiation (PCI) Collaborative Group. Standard-dose versus higher-dose prophylactic cranial irradiation (PCI) in patients with limited-stage small-cell lung cancer in complete remission after chemotherapy and thoracic radiotherapy (PCI 99-01, EORTC 22003-08004, RTOG 0212, and IFCT 99-01): a randomised clinical trial. Lancet Oncol. 2009 May;10(5):467-74. doi: 10.1016/S1470-2045(09)70101-9. Epub 2009 Apr 20. PMID 19386548
- [Background] Slotman BJ, Mauer ME, Bottomley A, Faivre-Finn C, Kramer GW, Rankin EM, Snee M, Hatton M, Postmus PE, Collette L, Senan S. Prophylactic cranial irradiation in extensive disease small-cell lung cancer: short-term health-related quality of life and patient reported symptoms: results of an international Phase III randomized controlled trial by the EORTC Radiation Oncology and Lung Cancer Groups. J Clin Oncol. 2009 Jan 1;27(1):78-84. doi: 10.1200/JCO.2008.17.0746. Epub 2008 Dec 1. PMID 19047288
- [Background] Sun A, Bae K, Gore EM, Movsas B, Wong SJ, Meyers CA, Bonner JA, Schild SE, Gaspar LE, Bogart JA, Werner-Wasik M, Choy H. Phase III trial of prophylactic cranial irradiation compared with observation in patients with locally advanced non-small-cell lung cancer: neurocognitive and quality-of-life analysis. J Clin Oncol. 2011 Jan 20;29(3):279-86. doi: 10.1200/JCO.2010.29.6053. Epub 2010 Dec 6. PMID 21135267
- [Background] Welzel G, Fleckenstein K, Schaefer J, Hermann B, Kraus-Tiefenbacher U, Mai SK, Wenz F. Memory function before and after whole brain radiotherapy in patients with and without brain metastases. Int J Radiat Oncol Biol Phys. 2008 Dec 1;72(5):1311-8. doi: 10.1016/j.ijrobp.2008.03.009. Epub 2008 Apr 28. PMID 18448270
- [Background] Auperin A, Arriagada R, Pignon JP, Le Pechoux C, Gregor A, Stephens RJ, Kristjansen PE, Johnson BE, Ueoka H, Wagner H, Aisner J. Prophylactic cranial irradiation for patients with small-cell lung cancer in complete remission. Prophylactic Cranial Irradiation Overview Collaborative Group. N Engl J Med. 1999 Aug 12;341(7):476-84. doi: 10.1056/NEJM199908123410703. PMID 10441603
- [Background] Bae K, Bruner DW, Baek S, Movsas B, Corn BW, Dignam JJ. Patterns of missing mini mental status exam (MMSE) in radiation therapy oncology group (RTOG) brain cancer trials. J Neurooncol. 2011 Nov;105(2):383-95. doi: 10.1007/s11060-011-0603-8. Epub 2011 May 21. PMID 21603964
- [Background] Kao J, Genden EM, Chen CT, Rivera M, Tong CC, Misiukiewicz K, Gupta V, Gurudutt V, Teng M, Packer SH. Phase 1 trial of concurrent erlotinib, celecoxib, and reirradiation for recurrent head and neck cancer. Cancer. 2011 Jul 15;117(14):3173-81. doi: 10.1002/cncr.25786. Epub 2011 Jan 18. PMID 21246519
- [Background] Metz JM, Smith D, Mick R, Lustig R, Mitchell J, Cherakuri M, Glatstein E, Hahn SM. A phase I study of topical Tempol for the prevention of alopecia induced by whole brain radiotherapy. Clin Cancer Res. 2004 Oct 1;10(19):6411-7. doi: 10.1158/1078-0432.CCR-04-0658. PMID 15475427
- [Background] Olsen EA. Investigative guidelines for alopecia areata. Dermatol Ther. 2011 May-Jun;24(3):311-9. doi: 10.1111/j.1529-8019.2011.01415.x. PMID 21689240